CLINICAL TRIAL: NCT06591637
Title: The Effects Of Fertility Supportive Behavior Education Based On Watson's Theory Of Human Care On Healthy Lifestyle Behaviors And İn Vitro Fertilization (IVF) Success İn Women With Primary Infertility
Brief Title: Fertility Supportive Behavior Education Based On Watson's Theory Of Human Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Duha Shaqalaih, PhD student, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1241/23
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Infertility, Female; IVF
Keywords: Fertility; Watson's Human Caring Theory; Lifestyle; Nursing Care
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group received fertility supportive behavior education based on Watson's Theory of Human Caring and was given a booklet titled 'Fertility-Supporting Health Training' at the onset of treatment. In addition to routine nursing care, the researcher provided detailed intervention and guidance regarding the booklet throughout the treatment period.
  Interventions: Behavioral: Fertility supportive behavior education based on Watson's Theory of Human Care; Procedure: Routine nursing care; Device: The booklet "Fertility-Supporting Health Training
- control group (Other): The control group received routine nursing care and was given a booklet titled 'Fertility-Supporting Health Training' at the onset of treatment, but the researcher did not provide any additional intervention or guidance regarding the booklet.
  Interventions: Procedure: Routine nursing care; Device: The booklet "Fertility-Supporting Health Training

INTERVENTIONS:
Behavioral: Fertility supportive behavior education based on Watson's Theory of Human Care — In this study, Watson's Theory of Human Caring guided the development of a care framework and nursing intervention for women with infertility. The researchers adapted the theory and focused on six of the ten carative factors : 1) Adopting values of humanity and devotion; 4) Developing supportive care relationships; 6) Using problem-solving methods for informed decisions; 7) Tailoring teaching to individual needs; 8) Creating a comfortable, peaceful environment; 9) Assisting with basic needs. The nursing care program, integrated with IVF treatments (14-18 days), involved four transpersonal interviews lasting 45-90 minutes each. These interviews were recorded in notes, used to individualize future sessions. The approach included active listening, empathy, and support, with participants encouraged to keep diaries for discussion. Communication was maintained in person, by phone, or email.
  Arms: intervention group
Procedure: Routine nursing care — Routine nursing care during IVF treatment includes:
  Pre-Treatment Counseling: Providing information and addressing patient questions.
  Monitoring and Assessment: Regular checks of health, hormone levels, and ovarian function.
  Medication Administration: Giving prescribed fertility drugs and other medications.
  Assisting with Procedures: Preparing and assisting with egg retrieval and embryo transfer.
  Emotional Support: Offering emotional and psychological support. Education: Instructing on medication use, self-care, and recognizing complications.
  Follow-Up Care: Scheduling and managing follow-up appointments to monitor progress
Device: The booklet "Fertility-Supporting Health Training — This booklet was prepared in line with the relevant literature and contained educational content aimed at improving healthy lifestyle behaviours . The training booklet included information on the effects of factors such as obesity, weakness, exposure to environmentally harmful substances, smoking and caffeine use on fertility and the methods of coping with these factors. In addition, information on how to use proper nutrition, develop exercise habits and cope with stress was provided. The booklet was distributed to the women at at the onset of the study.

SUMMARY:
Infertile individuals frequently attempt behavioral changes to enhance the effectiveness of their treatment and improve fertility outcomes. Consequently, this study was designed to assess the impact of fertility supportive behavior education, grounded in Watson's Human Care Theory, on healthy lifestyle behaviors and the success rates of in vitro fertilization (IVF) in women with primary infertility

ELIGIBILITY:
Inclusion Criteria:

* Women have a diagnosis of primary infertility.
* Women over the age of 18 and under the age of 32.
* Women able to read and write in Arabic.
* The cause of infertility must be a male factor.
* Women who are undergoing assisted reproductive techniques, specifically İn Vitro Fertilization-Intracytoplasmatic Sperm Injection.
* Women using the same drugs and protocols for IVF treatment.
* Only women who receive a fresh embryo transfer during their IVF treatment included in the study.

Exclusion Criteria:

* Women who have problems with understanding or perception
* The presence of tubal, uterine or other infertility factors in women
* Women undergoing a frozen embryo transfer as part of their IVF treatment
* Women whose pregnancies do not continue or who are diagnosed with a fetal anomaly by the time the healthy lifestyle behaviors scale is re-administered after 3 months excluded from the study.

Ages: 18 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The Health-Promoting Lifestyle Profile II instrument | Both groups completed a Health-Promoting Lifestyle Profile instrument and pre-test measures, at the onset of the study. At the end of treatment after embryo transfer they were administered test measures.After 3 months were administered posttest measure
  The Health-Promoting Lifestyle Profile II (HPLP-II) is a widely-used instrument for evaluation of health behaviour which has been validated in multiple studies. Based on Pender's Health Promotion Model, it conceptualises an individual's health-promoting lifestyle in terms of the following dimensions; health responsibility, physical activity, nutrition, spiritual growth, interpersonal relations and stress management.

SECONDARY OUTCOMES:
A quantitative human chorionic gonadotropin (HCG or hCG) blood test | 14 days after embryo transfer
  A quantitative human chorionic gonadotropin (HCG or hCG) blood test measures the specific level of HCG in the blood. HCG is a hormone produced in the body during pregnancy.
  Results are given in milli-international units per milliliter (mUI/mL).
  Normal levels are found in:
  Non-pregnant women: less than 5 milli-international units per milliliter Healthy men: less than 2 milli-international units per milliliter

CONTACTS AND LOCATIONS:
Locations (1):
- Albasma a private IVF center, Gaza, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No